CLINICAL TRIAL: NCT06801509
Title: A Randomized, Double-blind, Controlled Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the Recombinant Herpes Zoster Vaccine in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Recombinant Herpes Zoster Vaccine
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCTV04C-X201
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-Dose Vaccine Group (Experimental)
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (SCTV04C) Low-Dose
- High-Dose Vaccine Group (Experimental)
  Interventions: Biological: Recombinant Herpes Zoster Vaccine (SCTV04C) High-Dose
- Placebo Group (Placebo Comparator)
  Interventions: Biological: Placebo control: Saline
- Shingrix® Group (Active Comparator)
  Interventions: Biological: Shingrix®
- Ganwei® Group (Active Comparator): Herpes zoster vaccine, live; Changchun BCHT
  Interventions: Biological: Ganwei®

INTERVENTIONS:
Biological: Recombinant Herpes Zoster Vaccine (SCTV04C) Low-Dose — Route of vaccination: intramuscular injection into the lateral deltoid of the upper arm; Immunization procedure: 2 doses, 60 days apart;
  Arms: Low-Dose Vaccine Group
Biological: Recombinant Herpes Zoster Vaccine (SCTV04C) High-Dose — Route of vaccination: intramuscular injection into the lateral deltoid of the upper arm; Immunization procedure: 2 doses, 60 days apart;
  Arms: High-Dose Vaccine Group
Biological: Placebo control: Saline — The placebo in this study is 0.9% sodium chloride (normal saline) injection; Immunization procedure: 2 doses, 60 days apart;
  Arms: Placebo Group
Biological: Shingrix® — Route of vaccination: intramuscular injection into the lateral deltoid of the upper arm; Dosage of vaccination: 50 μg; Immunization procedure: 2 doses, 60 days apart
  Arms: Shingrix® Group
Biological: Ganwei® — Route of vaccination: subcutaneous injection into the lateral deltoid of the upper arm; Dosage of vaccination: 0.5 mL; Immunization procedure: saline will be administered at Day 0, and Ganwei® will be administered at Day 60；
  Arms: Ganwei® Group

SUMMARY:
The purposes of the study are to evaluate the Safety, Tolerability, and Immunogenicity of different dose levels of recombinant herpes zoster vaccine with 2 doses 60 days apart in healthy subjects aged 40 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 40 years of age;
2. The subject can and fully understand the trial procedures and voluntarily sign the ICF;
3. The subject is in a healthy state or has stable underlying diseases according to investigator's assessment based on medical history and related physical examination results;
4. The subject can comply with the requirements of the protocol;
5. The axillary temperature of the subject is < 37.0℃ on the day of enrollment;
6. Fertile men and women with childbearing potential voluntarily agree to take effective contraceptive measures from the first vaccination to at least 90 days after the last dose of study vaccines.

Exclusion Criteria:

1. History of herpes zoster before enrollment, or close contact with a varicella/herpes zoster patient within 30 days prior to enrollment;
2. Previous vaccination against herpes zoster and varicella (including vaccines that have been registered or under clinical research);
3. Allergic to any component of the study vaccine, or history of severe allergy to any vaccination, such as anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, local allergic necrosis reaction, angioneurotic edema, etc.
4. History or family history of convulsions, epilepsy, and psychiatric disorders;
5. Suffering from serious chronic diseases or in the active stage of chronic diseases, which are evaluated by the investigator to affect the trial observation, including but not limited to myocardial infarction, severe arrhythmia, unstable angina, hypertension that cannot be controlled after drug treatment (subjects 40-59 years of age have systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, and subjects ≥60 years of age have systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg), diabetes with severe complications, cancer or precancerous lesions, and other serious cerebrovascular diseases, heart disease, respiratory diseases, liver and kidney diseases, and thyroid diseases;
6. Primary or secondary immunosuppressive condition, or diagnosed with primary or acquired immunodeficiency disease, human immunodeficiency virus (HIV) infection, etc.
7. History of thrombocytopenia or other coagulation disorders, which may cause contraindications for intramuscular injection and venous blood collection;
8. Fever (axillary temperature ≥37.3℃) within 3 days before enrollment or systemic antibiotic or antiviral treatment within 7 days;
9. Use of antipyretic analgesics or other drugs with antipyretic and analgesic effects, such as acetaminophen and ibuprofen, within 72 h before vaccination.
10. Abnormal laboratory test (blood routine, blood biochemistry, urine routine) results that are outside the reference range and clinically significant (only apply to Phase I);
11. Those who are pregnant (positive urine pregnancy test) or breast-feeding, or those who plan to become pregnant during the study period;
12. Long-term or high-dose corticosteroid therapy (duration ≥15 days, or dose ≥1 mg/kg/ day of prednisone or equivalent doses of other corticosteroids), or other immunosuppressive and cytotoxic therapy within 90 days prior to vaccination. Short-term or topical use (such as ointments, eye drops, inhalants, intra-articular medications or nasal sprays) of glucocorticoids is permitted;
13. Vaccination with non-attenuated vaccines within 14 days before the first dose of study vaccines, or with live-attenuated vaccines within 28 days before the first dose of study vaccines;
14. Participation in other clinical trials (drug or vaccine) within 30 days preceding the first dose of study vaccines or planning to participate in other clinical trials before this clinical study is completed;
15. Asplenia or functional asplenia;
16. Those who are known to have been diagnosed or currently have an infectious disease, including hepatitis B, hepatitis C, syphilis or AIDS;
17. Those who have any acute illness or acute onset of chronic illness within 72 hours before the first dose of vaccination;
18. Those who have received blood or blood-related products, including immunoglobulins, within 3 months before the first dose of vaccination, or have planned to use them during the study period;
19. Subjects deemed by the investigator to have other conditions that render them ineligible to participate in this study, which include but are not limited to those who are incapable of participating in follow-up visits based on the protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
phase 1: Incidence and intensity of solicited adverse events (AEs) | within 14 days after each vaccination
phase 1: Incidence and intensity of unsolicited AEs | within 30 days after each vaccination
phase 2: Geometric mean concentration (GMC) and seroconversion rate of antigen-specific antibody | at 30 days after full vaccination

SECONDARY OUTCOMES:
phase 1: Geometric mean titer (GMT)/ GMC, Geometric mean fold increase (GMI), and seroconversion rate of antigen-, and VZV-specific antibody | at 30 days after the first vaccination, before the second vaccination, and at 30 days after full vaccination
phase 1:Frequency and response rate of CD4+ T cells with antigen-specific TNF-α and/or IFN-γ and/or IL-2 and/or CD40L secretion/expression as determined by intracellular cytokine staining (ICS) | at 30 days after the first vaccination, before the second vaccination, and at 30 days after full vaccination
phase 1: Incidence of Serious adverse events (SAEs) and Adverse events of special interest (AESIs) | during the study (from the first vaccination to 12 months after full vaccination)
phase 1: Incidence and intensity of abnormal laboratory tests indicators | 3 days after each vaccination
phase 2: GMI of antigen-specific antibody | at 30 days after full vaccination
phase 2: GMC, GMI, and seroconversion rate of antigen-specific antibody | before the second vaccination, and at 6 months, 12 months and 24 months after full vaccination
phase 2: GMT/GMC, GMI, and seroconversion rate of VZV-specific antibody | before the second vaccination, and at 30 days, 6 months, 12 months and 24 months after full vaccination
phase 2: Frequencies and response rate of CD4+ T cells with antigen-specific TNF-α and/or IFN-γ and/or IL-2 and/or CD40L secretion/expression as determined by ICS | before the second vaccination, and at 30 days, 6 months, 12 months and 24 months after full vaccination
phase 2: Incidence and intensity of solicited AEs | within 14 days after each vaccination
phase 2: Incidence and intensity of unsolicited AEs | within 30 days after each vaccination
phase 2: Incidence of SAEs and AESIs | from the first vaccination to 12 months after full vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Dazhu CDC, Dazhou, Sichuan, China